CLINICAL TRIAL: NCT01741857
Title: Phase I/II: Umbilical Cord Derived Mesenchymal Stem Cells Transplantation For Active And Refractory Systemic Lupus Erythematosus
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cells Transplantation for Active and Refractory Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Lingyun Sun, Department of Rheumatology and Immunology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJGLYY005
Record Dates: First submitted 2012-11-26; First posted 2012-12-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2012-10

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- human umbilical cord derived MSC (Experimental): human umbilical cord derived MSC transplantation for SLE
  Interventions: Biological: human umbilical cord derived MSC transplantation for SLE

INTERVENTIONS:
Biological: human umbilical cord derived MSC transplantation for SLE
  Other Names: Allogenic MSC derived from umbilical cord

SUMMARY:
This study will explore safety and efficacy of allogeneic umbilical cord (UC) derived mesenchymal stem cells transplantation (MSCT) to treat patients with active and refractory systemic lupus erythematosus (SLE) who have been resistant to multiple standard treatments. The underlying hypothesis is that the active SLE condition is caused by an abnormal immune homeostasis that can be restored by MSCT.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. All patients fulfilled the American College of Rheumatology (ACR) criteria of SLE, man or woman aged from 15 to 70 years old, SLEDAI≥8;
2. Lupus nephritis with 24h urine protein≥1g;
3. Refractory disease as determined by failure of the following regimens:

   Trial of corticosteroids (oral prednisone more than 20 mg/day); Trial of cyclophosphamide 0.4 ~ 0.6 / m2 every two weeks for six months, or other immunosuppressive drugs, such as mycophenolate mofetil 2 g / day, for three months;
4. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital;
5. Willing to use contraception throughout the study and for 12 months following treatment

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the American College of Rheumatology (ACR) criteria of SLE, man or woman aged from 15 to 60 years old, SLEDAI≥8;
* Lupus nephritis with 24h urine protein≥1g;
* Refractory disease as determined by failure of the following regimens:

Trial of corticosteroids (oral prednisone more than 20 mg/day); Trial of cyclophosphamide 0.4 ~ 0.6 / m2 every two weeks for six months, or other immunosuppressive drugs, such as mycophenolate mofetil 2 g / day, for three months;

* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital;
* Willing to use contraception throughout the study and for 12 months following treatment

Exclusion Criteria:

* Abnormal liver function (ALT higher than 3 times the normal value);
* End-stage renal failure;
* Severe heart and pulmonary failure, or other important organs damage;
* Uncontrolled infections
* Pregnant or breast feeding women, male or female who intended to recent pregnancy

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
British Isles Lupus Assessment Group score (BILAG) | up to 12 months

SECONDARY OUTCOMES:
Lupus serology (Alb, ANA, dsDNA, C3, C4) | pre-MSC transplantation, 1, 3, 6 and 12 months post MSC transplantation
Renal function (GFR, Blood Urea Nitrogen, urinalysis) | pre-MSC transplantation, 1, 3, 6 and 12 months post MSC transplantation (for GFR assessed at baseline and 12 months after MSCT)

CONTACTS AND LOCATIONS:
Overall Officials: Lingyun Sun, MD, PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Sun L, Akiyama K, Zhang H, Yamaza T, Hou Y, Zhao S, Xu T, Le A, Shi S. Mesenchymal stem cell transplantation reverses multiorgan dysfunction in systemic lupus erythematosus mice and humans. Stem Cells. 2009 Jun;27(6):1421-32. doi: 10.1002/stem.68. PMID 19489103
- [Background] Sun L, Wang D, Liang J, Zhang H, Feng X, Wang H, Hua B, Liu B, Ye S, Hu X, Xu W, Zeng X, Hou Y, Gilkeson GS, Silver RM, Lu L, Shi S. Umbilical cord mesenchymal stem cell transplantation in severe and refractory systemic lupus erythematosus. Arthritis Rheum. 2010 Aug;62(8):2467-75. doi: 10.1002/art.27548. PMID 20506343
- [Background] Liang J, Gu F, Wang H, Hua B, Hou Y, Shi S, Lu L, Sun L. Mesenchymal stem cell transplantation for diffuse alveolar hemorrhage in SLE. Nat Rev Rheumatol. 2010 Aug;6(8):486-9. doi: 10.1038/nrrheum.2010.80. Epub 2010 Jun 1. PMID 20517294
- [Background] Liang J, Zhang H, Hua B, Wang H, Lu L, Shi S, Hou Y, Zeng X, Gilkeson GS, Sun L. Allogenic mesenchymal stem cells transplantation in refractory systemic lupus erythematosus: a pilot clinical study. Ann Rheum Dis. 2010 Aug;69(8):1423-9. doi: 10.1136/ard.2009.123463. PMID 20650877
- [Background] Zhang H, Zeng X, Sun L. Allogenic bone-marrow-derived mesenchymal stem cells transplantation as a novel therapy for systemic lupus erythematosus. Expert Opin Biol Ther. 2010 May;10(5):701-9. doi: 10.1517/14712591003769816. PMID 20345339
- [Background] Shi D, Wang D, Li X, Zhang H, Che N, Lu Z, Sun L. Allogeneic transplantation of umbilical cord-derived mesenchymal stem cells for diffuse alveolar hemorrhage in systemic lupus erythematosus. Clin Rheumatol. 2012 May;31(5):841-6. doi: 10.1007/s10067-012-1943-2. PMID 22302582
- [Background] Che N, Li X, Zhou S, Liu R, Shi D, Lu L, Sun L. Umbilical cord mesenchymal stem cells suppress B-cell proliferation and differentiation. Cell Immunol. 2012;274(1-2):46-53. doi: 10.1016/j.cellimm.2012.02.004. Epub 2012 Feb 23. PMID 22414555
- [Background] Wang D, Akiyama K, Zhang H, Yamaza T, Li X, Feng X, Wang H, Hua B, Liu B, Xu H, Chen W, Shi S, Sun L. Double allogenic mesenchymal stem cells transplantations could not enhance therapeutic effect compared with single transplantation in systemic lupus erythematosus. Clin Dev Immunol. 2012;2012:273291. doi: 10.1155/2012/273291. Epub 2012 Jul 9. PMID 22829849
- [Derived] Li Z, Wang R, Wang D, Zhang S, Song H, Ding S, Zhu Y, Wen X, Li H, Chen H, Liu S, Sun L. Circulating miR-320b Contributes to CD4+ T-Cell Proliferation in Systemic Lupus Erythematosus via MAP3K1. J Immunol Res. 2023 Oct 26;2023:6696967. doi: 10.1155/2023/6696967. eCollection 2023. PMID 37928434
- [Derived] Wang D, Feng X, Lu L, Konkel JE, Zhang H, Chen Z, Li X, Gao X, Lu L, Shi S, Chen W, Sun L. A CD8 T cell/indoleamine 2,3-dioxygenase axis is required for mesenchymal stem cell suppression of human systemic lupus erythematosus. Arthritis Rheumatol. 2014 Aug;66(8):2234-45. doi: 10.1002/art.38674. PMID 24756936
- [Derived] Wang D, Li J, Zhang Y, Zhang M, Chen J, Li X, Hu X, Jiang S, Shi S, Sun L. Umbilical cord mesenchymal stem cell transplantation in active and refractory systemic lupus erythematosus: a multicenter clinical study. Arthritis Res Ther. 2014 Mar 25;16(2):R79. doi: 10.1186/ar4520. PMID 24661633